CLINICAL TRIAL: NCT06649006
Title: A Phase 1b Open-label Study to Investigate Safety, Tolerability and Pharmacokinetics of Intravenous Blinatumomab in Japanese Adult Subjects With Newly Diagnosed Philadelphia-negative B-precursor Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Study to Investigate Intravenous Blinatumomab in Japanese Adult Participants With Newly Diagnosed Philadelphia-negative B-precursor Acute Lymphoblastic Leukemia (B-ALL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230258
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: B-precursor Acute Lymphoblastic Leukemia
Keywords: Leukemia; Blincyto®; Blinatumomab; B-precursor Acute Lymphoblastic Leukemia; B-ALL
MeSH Terms: conditions — Leukemia | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab (Experimental): Participants affected by B-ALL will receive blinatumomab as an intravenous (IV) infusion.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — IV infusion
  Other Names: Blincyto®

SUMMARY:
The main objective of the study is to evaluate safety and tolerability of blinatumomab in adult Japanese participants with newly diagnosed B-ALL.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult participants ≥ 18 years and ≤ 70 years at enrollment.
* Participant should have newly diagnosed B-cell precursor (BCP)
* Philadelphia-negative ALL in CR/CRh after induction/consolidation therapy with any MRD (+ or -).
* CR/CRh as defined in Section 11.10, Appendix 10 after induction and at any time during consolidation chemotherapy with ALL MRD2008/2019/2023 protocol regimen or 3 blocks of Hyper-CVAD.
* Bone marrow function as defined below:

  * Absolute neutrophil count (ANC) (Neutrophils) ≥500/μL
  * Platelets ≥50.000/μL (transfusion permitted)
* Adequate renal and hepatic function:

  * Total bilirubin (TBL) ≤ 2.0 x upper limit of normal (ULN) (ULN; unless Gilbert's Disease or if liver involvement with leukemia)
  * Creatinine clearance ≥50 mL/min/1.73 m^2
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 2.

Exclusion Criteria:

Disease Related

* Current infiltration of cerebrospinal fluid (CSF) by ALL. If screening CSF demonstrates leukemic blasts, participants must receive intrathecal treatment and demonstrate negative CSF before enrollment and starting blinatumomab infusion.
* Immunotherapy (eg, rituximab, alemtuzumab) within 4 weeks before start of protocol-specified therapy.

Other Medical Conditions

* History of relevant central nervous system (CNS) pathology or current relevant CNS pathology (e.g., seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, or coordination or movement disorders).
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement.
* Active uncontrolled infection requiring therapy.
* History of other malignancy within the past 3 years, with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.

Prior/Concomitant Therapy

* Systemic cancer chemotherapy within 2 weeks prior to study treatment (except for intrathecal prophylaxis)
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus. In Japan, follow the JSH Guidelines for the Management of Hepatitis B Virus Infection version 4 (The Japan Society of Hepatology, 2022) for the screening of Hepatis B virus infection.
* Radiotherapy within 4 weeks prior to study treatment.

Prior/Concurrent Clinical Study Experience

• Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). This does not apply to other investigational procedures or participation in observational research studies while participating in this study are excluded.

Other Exclusions

* Participants of childbearing potential unwilling to use protocol-specified method of contraception during treatment and for an additional 48 hours after the last dose of blinatumomab.
* Participants who are breastfeeding or who plan to breastfeed while on study through 48 hours after the last dose of blinatumomab.
* Participants planning to become pregnant or donate eggs while on study through 48 hours after the last dose of blinatumomab.
* Participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive urine or serum pregnancy test.
* Participant has known hypersensitivity to blinatumomab or to any component of the product formulation.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety, or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately 31 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. A serious AE (SAE) is defined as any untoward medical occurrence that is: immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect.
Number of Participants Experiencing Adverse Events of Interest (EOI) | Up to 31 weeks

SECONDARY OUTCOMES:
Steady-state Concentration (Css) of Blinatumomab | Day 1 pre-dose, 2 and 6 hours post-dose on Day 1, Day 2, Day 3, Day 29
Clearance (CL) of Blinatumomab | Day 1 pre-dose, 2 and 6 hours post-dose on Day 1, Day 2, Day 3, Day 29
Number of Participants Achieving Minimal Residual Disease (MRD) After Each Cycle of Blinatumomab | Cycles 1-4: Day 29 (each cycle is 6 weeks)
Number of Participants Achieving Hematologic Complete Remission (CR) | Cycles 1-4: Day 29 (each cycle is 6 weeks)
Number of Participants Achieving Hematologic CR with Partial Peripheral Count Recovery (CRh) | Cycles 1-4: Day 29 (each cycle is 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- Japan (6):
  - Akita University Hospital, Akita, Akita
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yamagata University Hospital, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com